CLINICAL TRIAL: NCT04625985
Title: Adaptive Study to Demonstrate Efficacy and Safety of Metformin Glycinate for the Treatment of Hospitalized Patients With Severe Acute Respiratory Syndrome Secondary to SARS-CoV-2. Randomized, Double-Blind, Phase IIIb
Brief Title: Metformin Glycinate, Treatment of Patients With COVID-19 and Severe Acute Respiratory Syndrome Secondary to SARS-CoV-2.
Acronym: DMMETCOV19-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIL-30000-II-20(2)
Record Dates: First submitted 2020-10-23; First posted 2020-11-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: SARS-COV 2; Severe acute respiratory syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Experimental: Metformin glycinate 620 mg bid (PO) for 14 days plus standard treatment Control group: placebo bid (PO) for 14 days plus standard treatment
  Comparator: Placebo Placebo pill bid (PO) for 14 days plus standard treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parallel Assignment Experimental and placebo tablets will have same physical appearance and medicine box will be identified by kit number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin glycinate (Experimental): 620 mg bid (PO) for 14 days plus standard treatment
  Interventions: Drug: Metformin Glycinate
- Placebo (Placebo Comparator): Placebo tablet bid (PO) for 14 days plus standard treatment
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin Glycinate — Participants randomized to metformin glycinate will take 620 mg bid (PO) for 14 days plus standard treatment
  Other Names: DMMET
  Arms: Metformin glycinate
Drug: Placebo oral tablet — Participants randomized to placebo will take a tablet bid (PO) for 14 days in plus standard treatment
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the metformin glycinate and standard treatment of the hospital in hospitalized patients with Severe Acute Respiratory Syndrome secondary to SARS-CoV2.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1 day screening period to determine eligibility for study entry. At day 0, patients who meet the eligibility requirements will be randomized in a double blind manner (participant and investigator) in a 1:1 ratio to metformin glycinate (620 mg, taken orally, twice daily) plus standard treatment or placebo (taken orally, twice daily) plus standard treatment, both for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Ability to understand and the willingness to sign a written informed consent document before any study procedure
3. Coronavirus infection, severe acute respiratory syndrome (SARS-CoV)-2 confirmed by the polymerase chain reaction (PCR) test ≤ 4 days before randomization.
4. Hospitalized
5. Radiographic evidence of pulmonary infiltrates

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment for COVID-19
2. Evidence of multi-organ failure
3. Require mechanical ventilation before randomization
4. Pregnant patients
5. Patients with kidney failure, cancer and among other conditions that due to their treatment and / or baseline condition, affect the distribution, bioavailability and elimination of the studied drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Viral load | Day 0 to Day 28 or patient discharge day
  Assess differences in SARS-CoV-2 viral load between participants that receive placebo vs metformin glycinate
consciousness level | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of consciousness level: alertness
temperature | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of axillary body temperature in °C: <37.2.
systolic blood pressure | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of systolic blood pressure in mmHg: >90.
Oxigen saturation | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of oxygen saturation in %: >90.
Heart rate | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of heart rate in beats per minute: <100 bpm.
respiratory rate | Day 0 to Day 28 or patient discharge day
  Clinical status assessed by measurement of respiratory rate in breaths per minute: <24 bpm,
Days of hospitalization | Day 0 to Day 28 or patient discharge day
  Assess length of hospitalization
Days of supplementary oxygen if applies | Day 0 to Day 28 or patient discharge day
  Assess length of supplementary oxygen
Days of supplementary mechanical ventilation | Day 0 to Day 28 or patient discharge day
  Assess length of mechanical ventilation

SECONDARY OUTCOMES:
Toxicity of study drug assessed by incidence of adverse events (grade 3 or 4) | Day 0 to Day 28 or patient discharge day
  Assess by incidence of Grade 3, Grade 4, and Serious Adverse Events (AEs)
Changes in laboratory test results | Day 0 to Day 28 or patient discharge day
  Changes in serum levels from security laboratories compared to baseline levels and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Silvia M Aguirre, MD, Principal Investigator — The American British Cowdray Medical Center. I.A.P.
Locations (1):
- The American British Cowdray Medical Center, I.A.P, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer M, Timper K, Radimerski T, Dembinski K, Frey DM, Zulewski H, Keller U, Muller B, Christ-Crain M, Grisouard J. Metformin induces glucose uptake in human preadipocyte-derived adipocytes from various fat depots. Diabetes Obes Metab. 2010 Apr;12(4):356-9. doi: 10.1111/j.1463-1326.2009.01169.x. PMID 20380657
- [Background] Cuthbertson J, Patterson S, O'Harte FP, Bell PM. Investigation of the effect of oral metformin on dipeptidylpeptidase-4 (DPP-4) activity in Type 2 diabetes. Diabet Med. 2009 Jun;26(6):649-54. doi: 10.1111/j.1464-5491.2009.02748.x. PMID 19538242
- [Result] Musi N, Hirshman MF, Nygren J, Svanfeldt M, Bavenholm P, Rooyackers O, Zhou G, Williamson JM, Ljunqvist O, Efendic S, Moller DE, Thorell A, Goodyear LJ. Metformin increases AMP-activated protein kinase activity in skeletal muscle of subjects with type 2 diabetes. Diabetes. 2002 Jul;51(7):2074-81. doi: 10.2337/diabetes.51.7.2074. PMID 12086935
- [Result] Shaw RJ, Lamia KA, Vasquez D, Koo SH, Bardeesy N, Depinho RA, Montminy M, Cantley LC. The kinase LKB1 mediates glucose homeostasis in liver and therapeutic effects of metformin. Science. 2005 Dec 9;310(5754):1642-6. doi: 10.1126/science.1120781. Epub 2005 Nov 24. PMID 16308421
- [Result] Detaille D, Guigas B, Leverve X, Wiernsperger N, Devos P. Obligatory role of membrane events in the regulatory effect of metformin on the respiratory chain function. Biochem Pharmacol. 2002 Apr 1;63(7):1259-72. doi: 10.1016/s0006-2952(02)00858-4. PMID 11960602
- [Result] Tamura Y, Watada H, Sato F, Kumashiro N, Sakurai Y, Hirose T, Tanaka Y, Kawamori R. Effects of metformin on peripheral insulin sensitivity and intracellular lipid contents in muscle and liver of overweight Japanese subjects. Diabetes Obes Metab. 2008 Sep;10(9):733-8. doi: 10.1111/j.1463-1326.2007.00801.x. Epub 2007 Oct 15. PMID 17941868
- [Result] Standeven KF, Ariens RA, Whitaker P, Ashcroft AE, Weisel JW, Grant PJ. The effect of dimethylbiguanide on thrombin activity, FXIII activation, fibrin polymerization, and fibrin clot formation. Diabetes. 2002 Jan;51(1):189-97. doi: 10.2337/diabetes.51.1.189. PMID 11756340
- [Result] Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Ramos-Zavala MG, Barrera-Duran C, Gonzalez-Canudas J. Effect of metformin glycinate on glycated hemoglobin A1C concentration and insulin sensitivity in drug-naive adult patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2012 Dec;14(12):1140-4. doi: 10.1089/dia.2012.0097. Epub 2012 Sep 13. PMID 22974412
- [Result] Jorge González Canudas, COMET GROUP Diabetes Efficacy and Safety of Metformin Glycinate vs. Metformin Hydrochloride in Metabolic Control and Inflammatory Mediators in Type 2 Diabetes Mellitus Patients. Diabetes 2019 Jun; 68(Supplement 1)
- [Result] Garza-Ocañas L, Tamez-de la O E, Iglesias-Chiesa J, Gonzalez Canudas J, Rivas-Ruiz R: Pharmacokinetics and gastrointestinal tolerability of DMMET 01 (glycinate of metformin): results of a prospective randomized trial in healthy volunteers [abstract]. Diabetes 2009;58(Suppl 1):A533